CLINICAL TRIAL: NCT05148962
Title: A Phase 1 Trial to Evaluate the Safety, Immunogenicity, and Reactogenicity of a Self-Amplifying mRNA Prophylactic Vaccine Boost Against SARS-CoV-2 in Previously Vaccinated Healthy Adults 18 Years and Older
Brief Title: Study of GRT-R910 COVID-19 Boost Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GO-009
Record Dates: First submitted 2021-12-03; First posted 2021-12-08 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 vaccine; Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — GRT-R910 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1: GRT-R910 10 µg, age ≥60 years (Receipt of AstraZeneca vaccine) (Experimental): Healthy participants of age ≥60 years received prime dose (on Day 1) of GRT-R910 10 microgram (µg) intramuscularly at least 2 months after receiving a first-generation COVID-19 (AstraZeneca) vaccine primary series. A subset of participants elected to receive a booster vaccination of GRT-R910 10 µg which was administered 113 days after the prime vaccination. Participants not receiving booster dose were followed for 12 months, and participants receiving booster dose were followed for 16 months.
  Interventions: Biological: GRT-R910
- Cohort 2: GRT-R910 30 µg, age ≥60 years (Receipt of AstraZeneca vaccine) (Experimental): Healthy participants of age ≥60 years received prime dose (on Day 1) of GRT-R910 30 µg intramuscularly at least 2 months after receiving a first-generation COVID-19 (AstraZeneca) vaccine primary series. A subset of participants elected to receive a booster vaccination of GRT-R910 10 µg, which was administered 113 days after the prime vaccination. Participants not receiving booster dose were followed for 12 months, and participants receiving booster dose were followed for 16 months.
  Interventions: Biological: GRT-R910
- Cohort 3: GRT-R910 10 µg, ≥60 years, (Receipt of AstraZeneca or Janssen COVID-19 vaccine) (Experimental): Healthy participants of age ≥60 years received two doses (Day 1 and Day 29) of GRT-R910 10 µg (homologous prime-boost), at least 2 months after receiving an adenoviral COVID-19 (AstraZeneca, Janssen) primary series vaccine. Participants were followed for 13 months.
  Interventions: Biological: GRT-R910
- Cohort 4: GRT-R910 10 µg, ≥60 years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 vaccine) (Experimental): Healthy participants of age ≥60 years received two doses (Day 1 and Day 29) of GRT-R910 10 µg (homologous prime-boost), at least 2 months after receiving a messenger ribonucleic acid (mRNA)-based COVID-19 (Pfizer/BioNTech, Moderna) primary series vaccine. Participants were followed for 13 months.
  Interventions: Biological: GRT-R910
- Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 vaccine) (Experimental): Healthy participants of age ≥18 to ≤59 years received two doses (Day 1 and Day 29) of GRT-R910 10 µg (homologous prime-boost), at least 2 months after receiving mRNA-based COVID-19 (Pfizer/BioNTech, Moderna) primary series vaccine. Participants were followed for 13 months.
  Interventions: Biological: GRT-R910

INTERVENTIONS:
Biological: GRT-R910 — Injection administered intramuscularly

SUMMARY:
The primary objective was to assess the safety and tolerability of 2 different doses (10 or 30 µg) of GRT-R910 when administered as a boost in healthy adults previously vaccinated with the AstraZeneca, Janssen/Johnson and Johnson, Moderna, or Pfizer/BioNTech Coronavirus disease 2019 (COVID-19) vaccines.

DETAILED DESCRIPTION:
This trial studied a self-amplifying messenger ribonucleic acid (samRNA) based vaccine (GRT-R910) in previously vaccinated adults (≥18 years). GRT-R910 uses a codon optimized, prefusion stabilized Spike (S) cassette with additional T cell epitopes (TCEs) covering multiple epitopes from non-spike proteins to safely drive strong, broad, and durable B and T cell immune responses to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2).

ELIGIBILITY:
Inclusion Criteria:

* For Cohorts 1 and 2, have received AstraZeneca's AZD1222 COVID-19 prime and boost vaccine (Covishield®, Vaxzevria®), with the last dose received at least 2 months or more prior to Day 1.
* For Cohort 3, have received a primary series of an adenoviral (AstraZeneca AZD1222 [Covishield®, Vaxzevria®] or Janssen [Janssen COVID-19 Vaccine]) COVID-19 vaccine (under emergency supply procedures or upon full approval and may have received booster doses of an authorized vaccine), with the last dose received at least 2 months or more prior to Day 1.
* For Cohorts 4 and 6, have received a primary series of an mRNA (Pfizer/BioNTech [Comirnaty®] or Moderna [Spikevax®]) COVID-19 vaccine (under emergency supply procedures or upon full approval and may have received booster doses of an authorized vaccine), with the last dose received at least 2 months or more prior to Day 1.
* Agree to refrain from blood donation during the course of the study.
* Women of childbearing potential (WOCBP)* must agree to avoid pregnancy and be willing to use a highly effective method of contraception** consistently for 30 days prior to the first study vaccine and for at least 60 days after the last study vaccine
* Male subjects of childbearing potential must agree to the use of condoms to ensure effective contraception with a female partner from the time of study vaccination until 3 months after vaccination. Male subjects agree to refrain from sperm donation from the time of first vaccination until 3 months after the last vaccination. Male subjects of childbearing potential are biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
* Plan to remain living in the area for the duration of the study.

Exclusion Criteria:

* History of prior confirmed COVID-19 (cohorts 1 and 2).
* History of prior confirmed (polymerase chain reaction [PCR] or antigen test positive) COVID-19 infection as confirmed by a diagnostic laboratory less than 16 weeks (112 days) prior to enrollment (Cohorts 3, 4, and 6).
* Positive for SARS-CoV-2 (N-specific) antibody testing and had a history of upper respiratory illness consistent with COVID-19 within the 112 days prior to enrollment (Cohorts 3, 4, and 6).
* Prior receipt of a SARS-CoV-2 vaccine other than AstraZeneca's AZD1222 (Covishield®, Vaxzevria®), JNJ-78436735, Pfizer/BioNTech (Comirnaty®), Moderna (Spikevax®), other approved or investigational adenovirus vectored vaccines, approved or investigational vaccines with a lipid nanoparticle (LNP) component, or any other approved or investigational vaccine likely to impact the interpretation of the trial data.
* On current treatment or prevention agents with activity against SARS-CoV-2.
* Participation in another research study involving receipt of an investigational product in the 60 days preceding enrollment or planned use during the study period.
* Receipt or planned receipt of any live, attenuated vaccine within 28 days before or after study vaccination.
* Receipt or planned receipt of any subunit or killed vaccine within 14 days before or after vaccination.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the planned administration of first study vaccination or at any time during the study.
* Breastfeeding, pregnant, or planning to become pregnant during the course of the study.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection with CD4+ T-cells < 400/mm3, asplenia, recurrent, severe infections and chronic (more than 14 continuous days) immunosuppressant medication within the past 6 months (inhaled, ophthalmic, and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including urticaria, respiratory difficulty or abdominal pain (or any immediate allergic reaction of any severity to polysorbate due to potential cross-reactive hypersensitivity with the PEG component of the vaccine).
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis, including but not limited to reaction to vaccination.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious ongoing, unstable psychiatric condition that in the opinion of the investigator would interfere with study participation.
* Bleeding disorder or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Suspected or known current alcohol abuse that in the opinion of the investigator would impede compliance with the protocol and schedules of assessments.
* Suspected or known current alcohol abuse that in the opinion of the investigator would impede compliance with the protocol and schedules of assessments. Suspected or known drug abuse in the 5 years preceding enrollment.
* Any other condition that in the opinion of the investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Martin, DO, Study Director — Gritstone bio, Inc.
Locations (3):
- United Kingdom (3):
  - University Hospitals Birmingham NHS, Birmingham
  - University Hospital of Leicester NHS Trust, Leicester
  - Manchester University, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer CD, Scallan CD, Kraemer Tardif LD, Kachura MA, Rappaport AR, Koralek DO, Uriel A, Gitlin L, Klein J, Davis MJ, Venkatraman H, Hart MG, Jaroslavsky JR, Kounlavouth S, Marrali M, Nganje CN, Bae K, Yan T, Leodones K, Egorova M, Hong SJ, Kuan J, Grappi S, Garbes P, Jooss K, Ustianowski A. GRT-R910: a self-amplifying mRNA SARS-CoV-2 vaccine boosts immunity for >/=6 months in previously-vaccinated older adults. Nat Commun. 2023 Jun 6;14(1):3274. doi: 10.1038/s41467-023-39053-9. PMID 37280238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled at 3 sites in United Kingdom. A total of 61 participants were screened and 45 participants were enrolled in 6 cohorts (Cohorts 1 to 6).
Pre-assignment Details: Of 45 enrolled participants, 1 participant was enrolled in Cohort 5; however, the sponsor decided to terminate this participant prior to the study vaccination and close the recruitment of Cohort 5. As a result, Cohort 5 was removed from the GO-009 study. Therefore, the results include participants enrolled in Cohorts 1, 2, 3, 4, and 6.
Groups:
- Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine): Healthy participants of age ≥60 years received prime dose (on Day 1) of GRT-R910 10 µg intramuscularly at least 2 months after receiving a first-generation COVID-19 (AstraZeneca) vaccine primary series. A subset of participants elected to receive a booster vaccination of GRT-R910 10 µg which was administered 113 days after the prime vaccination. Participants not receiving booster dose were followed for 12 months, and participants receiving booster dose were followed for 16 months.
Period: Overall Study
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Started | 11 | 8 | 10 | 12 | 3
Vaccinated | 10 | 7 | 10 | 10 | 3
Completed | 10 | 7 | 7 | 5 | 1
Not Completed | 1 | 1 | 3 | 7 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0
Not completed — Participant was early terminated per protocol | 0 | 0 | 3 | 5 | 2
Not completed — Miscellaneous | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Population (SAF) included all participants who received any dose of GRT-R910.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Total
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.61) | 66.7 (5.06) | 65.5 (3.95) | 73.5 (5.40) | 33.0 (11.36) | 66.1 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 4 | 2 | 19
  Male | 6 | 2 | 6 | 6 | 1 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 10 | 10 | 3 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 8 | 6 | 9 | 10 | 2 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Solicited Local Adverse Event (AE) Within 8 Days After the Injection of Prime Dose
Description: An AE was defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related in a participant or clinical investigation participant who administered a pharmaceutical product regardless of its causal relationship to the study treatment. Solicited local AEs included injection site pain, injection site tenderness, injection site erythema, injection site edema/induration. Solicited AEs (reactogenicity) were collected using a memory aid.
Time Frame: Within 8 Days After the Injection of Prime Dose on Day 1
Population: SAF population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
Participants | 8 | 6 | 10 | 10 | 3

2. Primary Outcome: Number of Participants With at Least One Solicited Local AE Within 8 Days After the Injection of Booster Dose
Description: as for outcome 1
Time Frame: Within 8 Days After the Injection of Booster Dose on Day 113 (Cohorts 1, 2); Within 8 Days After the Injection of Booster Dose on Day 29 (Cohorts 3, 4, 6)
Population: Participants in the SAF population who received booster dose and submitted any data for the solicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 6 | 4 | 8 | 7 | 3
Participants | 6 | 4 | 8 | 6 | 3

3. Primary Outcome: Number of Participants With at Least One Solicited Systemic AE Within 8 Days After the Injection of Prime Dose
Description: An AE was defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related in a participant or clinical investigation participant who administered a pharmaceutical product regardless of its causal relationship to the study treatment. Solicited systemic AEs included headache, fatigue, malaise, myalgia, arthralgia, nausea, fever, and chills. Solicited AEs (reactogenicity) were collected using a memory aid.
Time Frame: Within 8 Days After the Injection of Prime Dose on Day 1
Population: SAF population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
Participants | 8 | 7 | 10 | 9 | 3

4. Primary Outcome: Number of Participants With at Least One Solicited Systemic AE Within 8 Days After the Injection of Booster Dose
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Participants in the SAF population who received booster dose and submitted any data for the solicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 6 | 4 | 8 | 7 | 3
Participants | 4 | 4 | 8 | 6 | 3

5. Primary Outcome: Number of Participants With at Least One Unsolicited Treatment-emergent AEs (TEAEs) Within 28 Days After the Injection of Prime Dose
Description: An AE was defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related in a participant or clinical investigation participant who administered a pharmaceutical product regardless of its causal relationship to the study treatment. A TEAE was defined as any event not observed before the first vaccination or any event observed before the first vaccination that worsens in intensity or frequency after exposure.
Time Frame: Within 28 Days After the Injection of Prime Dose on Day 1
Population: SAF population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
Participants | 5 | 6 | 7 | 8 | 3

6. Primary Outcome: Number of Participants With at Least One Unsolicited TEAEs Within 28 Days After the Injection of Booster Dose
Description: as for outcome 5
Time Frame: Within 28 Days After the Injection of Booster Dose on Day 113 (Cohorts 1, 2); Within 8 Days After the Injection of Booster Dose on Day 29 (Cohorts 3, 4, 6)
Population: Participants in the SAF population who received booster dose were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 6 | 4 | 8 | 7 | 3
Participants | 4 | 4 | 4 | 4 | 2

7. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes at Day 8 in Participants Without Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in SAF population from Cohorts 1 and 2 who did not receive the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 4 | 3
10^9 cells per liter
  Basophils : Baseline | 0.033 (0.0150) | 0.017 (0.0153)
  Basophils : Change at Day 8 | -0.003 (0.0126) | -0.003 (0.0115)
  Eosinophils : Baseline | 0.185 (0.1420) | 0.137 (0.0874)
  Eosinophils : Change at Day 8 | 0.073 (0.1333) | -0.040 (0.0794)
  Lymphocytes : Baseline | 1.338 (0.7852) | 1.203 (0.8739)
  Lymphocytes : Change at Day 8 | -0.053 (0.2109) | -0.187 (0.5052)
  Monocytes : Baseline | 0.430 (0.1722) | 0.570 (0.1442)
  Monocytes : Change at Day 8 | -0.023 (0.1195) | 0.010 (0.0500)
  Neutrophils : Baseline | 3.170 (1.1786) | 5.057 (0.5036)
  Neutrophils : Change at Day 8 | -0.443 (0.9483) | -1.610 (0.9681)
  Platelets : Baseline | 199.8 (65.20) | 276.0 (53.86)
  Platelets : Change at Day 8 | -5.5 (19.49) | -39.0 (29.87)
  Leukocytes : Baseline | 5.15 (1.808) | 7.00 (0.794)
  Leukocytes : Change at Day 8 | -0.43 (1.348) | -1.83 (1.266)

8. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes at Day 8 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
10^9 cells per liter
  Basophils : Baseline | 0.040 (0.0126) | 0.063 (0.0359)
  Basophils : Change at Day 8 | -0.020 (0.0110) | -0.030 (0.0216)
  Eosinophils : Baseline | 0.128 (0.1783) | 0.143 (0.0846)
  Eosinophils : Change at Day 8 | 0.037 (0.0866) | -0.043 (0.0150)
  Lymphocytes : Baseline | 1.510 (0.3653) | 1.610 (0.3350)
  Lymphocytes : Change at Day 8 | 0.088 (0.1731) | -0.223 (0.1209)
  Monocytes : Baseline | 0.490 (0.1456) | 0.558 (0.2152)
  Monocytes : Change at Day 8 | -0.028 (0.0708) | -0.053 (0.0789)
  Neutrophils : Baseline | 5.205 (1.3505) | 4.003 (1.3023)
  Neutrophils : Change at Day 8 | -1.165 (0.8976) | -0.970 (1.0519)
  Platelets : Baseline | 269.0 (95.68) | 271.8 (21.36)
  Platelets : Change at Day 8 | -43.5 (54.70) | -26.5 (42.07)
  Leukocytes : Baseline | 7.37 (1.325) | 6.40 (1.679)
  Leukocytes : Change at Day 8 | -1.07 (0.954) | -1.35 (0.929)

9. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes at Day 120 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 120
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
10^9 cells per liter
  Basophils : Baseline | 0.040 (0.0126) | 0.063 (0.0359)
  Basophils : Change at Day 120 | -0.013 (0.0103) | -0.030 (0.0163)
  Eosinophils : Baseline | 0.128 (0.1783) | 0.143 (0.0846)
  Eosinophils : Change at Day 120 | 0.032 (0.0581) | -0.013 (0.0263)
  Lymphocytes : Baseline | 1.510 (0.3653) | 1.610 (0.3350)
  Lymphocytes : Change at Day 120 | 0.192 (0.1873) | -0.143 (0.1477)
  Monocytes : Baseline | 0.490 (0.1456) | 0.558 (0.2152)
  Monocytes : Change at Day 120 | -0.040 (0.0363) | -0.108 (0.1646)
  Neutrophils : Baseline | 5.205 (1.3505) | 4.003 (1.3023)
  Neutrophils : Change at Day 120 | -2.040 (0.8313) | -1.170 (0.3218)
  Platelets : Baseline | 269.0 (95.68) | 271.8 (21.36)
  Platelets : Change at Day 120 | -21.3 (36.79) | -31.5 (54.86)
  Leukocytes : Baseline | 7.37 (1.325) | 6.40 (1.679)
  Leukocytes : Change at Day 120 | -1.87 (0.898) | -1.50 (0.392)

10. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes at Day 8 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 3, 4 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
10^9 cells per liter
  Basophils : Baseline | 0.047 (0.0250) | 0.047 (0.0125) | 0.043 (0.0115)
  Basophils : Change at Day 8 | -0.020 (0.0176) | -0.022 (0.0132) | -0.023 (0.0058)
  Eosinophils : Baseline | 0.123 (0.1311) | 0.126 (0.0875) | 0.107 (0.0569)
  Eosinophils : Change at Day 8 | 0.022 (0.0721) | 0.009 (0.0493) | -0.047 (0.0289)
  Lymphocytes : Baseline | 1.574 (0.4610) | 1.639 (0.9816) | 1.507 (0.1793)
  Lymphocytes : Change at Day 8 | -0.006 (0.2913) | -0.170 (0.2732) | -0.293 (0.0306)
  Monocytes : Baseline | 0.481 (0.1194) | 0.508 (0.1160) | 0.373 (0.1464)
  Monocytes : Change at Day 8 | -0.066 (0.0929) | -0.131 (0.1058) | -0.120 (0.1323)
  Neutrophils : Baseline | 3.701 (1.4781) | 3.921 (0.7834) | 2.643 (0.6831)
  Neutrophils : Change at Day 8 | -0.645 (0.7103) | -1.041 (0.6897) | -0.920 (0.9885)
  Platelets : Baseline | 230.2 (30.53) | 249.4 (59.23) | 267.0 (23.58)
  Platelets : Change at Day 8 | 12.5 (41.25) | -20.3 (25.58) | -19.7 (70.32)
  Leukocytes : Baseline | 5.920 (1.7261) | 6.240 (1.2834) | 4.633 (0.7506)
  Leukocytes : Change at Day 8 | -0.650 (0.9058) | -1.350 (0.6042) | -1.367 (0.8963)

11. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets, Leukocytes at Day 37 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 37
Population: Participants in the SAF population from Cohorts 3, 4 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
10^9 cells per liter
  Basophils : Baseline | 0.047 (0.0250) | 0.047 (0.0125) | 0.043 (0.0115)
  Basophils : Change at Day 37 | -0.013 (0.0116) | -0.014 (0.0117) | -0.017 (0.0115)
  Eosinophils : Baseline | 0.123 (0.1311) | 0.126 (0.0875) | 0.107 (0.0569)
  Eosinophils : Change at Day 37 | 0.013 (0.0523) | 0.001 (0.0669) | -0.033 (0.0153)
  Lymphocytes : Baseline | 1.574 (0.4610) | 1.639 (0.9816) | 1.507 (0.1793)
  Lymphocytes : Change at Day 37 | 0.021 (0.3380) | -0.140 (0.3636) | -0.253 (0.1343)
  Monocytes : Baseline | 0.481 (0.1194) | 0.508 (0.1160) | 0.373 (0.1464)
  Monocytes : Change at Day 37 | 0.033 (0.1585) | -0.107 (0.1846) | -0.030 (0.1044)
  Neutrophils : Baseline | 3.701 (1.4781) | 3.921 (0.7834) | 2.643 (0.6831)
  Neutrophils : Change at Day 37 | -0.136 (0.8558) | -0.125 (0.7983) | 0.000 (1.4504)
  Platelets : Baseline | 230.2 (30.53) | 249.4 (59.23) | 267.0 (23.58)
  Platelets : Change at Day 37 | 37.4 (65.25) | -4.5 (21.18) | 13.3 (60.68)
  Leukocytes : Baseline | 5.920 (1.7261) | 6.240 (1.2834) | 4.633 (0.7506)
  Leukocytes : Change at Day 37 | -0.070 (0.9900) | -0.390 (0.8556) | -0.280 (1.4153)

12. Primary Outcome: Change From Baseline in Hemoglobin at Day 8 in Participants Without Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who did not receive the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 4 | 3
g/L
  Hemoglobin : Baseline | 131.5 (12.58) | 136.7 (11.85)
  Hemoglobin : Change at Day 8 | -3.8 (3.50) | -4.0 (1.73)

13. Primary Outcome: Change From Baseline in Hemoglobin at Day 8 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
g/L
  Hemoglobin : Baseline | 137.8 (13.01) | 144.8 (7.97)
  Hemoglobin : Change at Day 8 | -5.5 (5.24) | -7.0 (10.10)

14. Primary Outcome: Change From Baseline in Hemoglobin at Day 120 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 120
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
g/L
  Hemoglobin : Baseline | 137.8 (13.01) | 144.8 (7.97)
  Hemoglobin : Change at Day 120 | -4.8 (4.54) | -5.3 (2.75)

15. Primary Outcome: Change From Baseline in Hemoglobin at Day 8 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 3, 4 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
g/L
  Hemoglobin : Baseline | 136.3 (9.25) | 139.0 (8.69) | 130.3 (6.03)
  Hemoglobin : Change at Day 8 | -5.9 (3.25) | -4.8 (5.45) | -5.7 (6.35)

16. Primary Outcome: Change From Baseline in Hemoglobin at Day 37 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 37
Population: Participants in the SAF population from Cohorts 3, 4 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
g/L
  Hemoglobin : Baseline | 136.3 (9.25) | 139.0 (8.69) | 130.3 (6.03)
  Hemoglobin : Change at Day 37 | -8.0 (4.62) | -6.6 (4.53) | -11.0 (6.08)

17. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at Day 8 in Participants Without Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who did not receive the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: International Units Per Liter (IU/L)
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 4 | 3
International Units Per Liter (IU/L)
  Alkaline Phosphatase : Baseline | 75.0 (14.63) | 81.3 (24.01)
  Alkaline Phosphatase : Change at Day 8 | 4.8 (13.35) | 1.7 (8.33)
  Alanine Aminotransferase : Baseline | 22.3 (7.63) | 17.3 (3.51)
  Alanine Aminotransferase : Change at Day 8 | 11.8 (29.93) | 38.7 (39.32)
  Aspartate Aminotransferase : Baseline | 24.5 (5.20) | 18.7 (2.89)
  Aspartate Aminotransferase : Change at Day 8 | 5.3 (11.35) | 14.7 (10.97)

18. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at Day 8 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose and who had available data were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
IU/L
  Alkaline Phosphatase : Baseline | 82.5 (20.50) | 67.5 (35.75)
  Alkaline Phosphatase : Change at Day 8 | 4.8 (22.97) | -12.5 (8.96)
  Alanine Aminotransferase : Baseline | 25.5 (13.34) | 18.3 (9.39)
  Alanine Aminotransferase : Change at Day 8 | 2.5 (14.54) | 3.5 (8.66)
  Aspartate Aminotransferase : Baseline | 23.5 (8.38) | 18.8 (1.50)
  Aspartate Aminotransferase : Change at Day 8: number analyzed (Participants) | 5 | 4
  Aspartate Aminotransferase : Change at Day 8 | 0.6 (6.66) | 3.0 (4.08)

19. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at Day 120 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 120
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
IU/L
  Alkaline Phosphatase : Baseline | 82.5 (20.50) | 67.5 (35.75)
  Alkaline Phosphatase : Change at Day 120 | -2.8 (18.65) | -13.5 (10.41)
  Alanine Aminotransferase : Baseline | 25.5 (13.34) | 18.3 (9.39)
  Alanine Aminotransferase : Change at Day 120 | -4.0 (11.03) | 4.3 (5.68)
  Aspartate Aminotransferase : Baseline | 23.5 (8.38) | 18.8 (1.50)
  Aspartate Aminotransferase : Change at Day 120: number analyzed (Participants) | 4 | 3
  Aspartate Aminotransferase : Change at Day 120 | -0.8 (4.50) | 1.0 (3.46)

20. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at Day 8 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 8
Population: Participants in SAF population from Cohorts 3, 4, and 6 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
IU/L
  Alkaline Phosphatase : Baseline | 75.0 (19.96) | 83.9 (20.56) | 58.7 (6.81)
  Alkaline Phosphatase : Change at Day 8 | 7.7 (10.67) | -6.8 (13.10) | -4.7 (1.15)
  Alanine Aminotransferase : Baseline | 25.6 (8.62) | 25.1 (9.42) | 14.3 (5.51)
  Alanine Aminotransferase : Change at Day 8 | -0.4 (5.17) | 7.2 (15.10) | 10.0 (14.73)
  Aspartate Aminotransferase : Baseline | 25.2 (6.27) | 26.1 (5.71) | 21.5 (2.12)
  Aspartate Aminotransferase : Change at Day 8: number analyzed (Participants) | 10 | 9 | 2
  Aspartate Aminotransferase : Change at Day 8 | -0.1 (4.51) | 1.9 (8.55) | 1.5 (9.19)

21. Primary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, and Aspartate Aminotransferase at Day 37 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 37
Population: Participants in SAF population from Cohorts 3, 4, and 6 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
IU/L
  Alkaline Phosphatase : Baseline | 75.0 (19.96) | 83.9 (20.56) | 58.7 (6.81)
  Alkaline Phosphatase : Change at Day 37 | -7.9 (8.13) | 0.2 (11.44) | -1.7 (1.15)
  Alanine Aminotransferase : Baseline | 25.6 (8.62) | 25.1 (9.42) | 14.3 (5.51)
  Alanine Aminotransferase : Change at Day 37 | 0.7 (7.83) | 3.2 (6.92) | 2.7 (0.58)
  Aspartate Aminotransferase : Baseline: number analyzed (Participants) | 10 | 9 | 2
  Aspartate Aminotransferase : Baseline | 25.2 (6.27) | 26.1 (5.71) | 21.5 (2.12)
  Aspartate Aminotransferase : Change at Day 37: number analyzed (Participants) | 9 | 7 | 1
  Aspartate Aminotransferase : Change at Day 37 | 1.9 (7.04) | 3.1 (8.61) | -1.0

22. Primary Outcome: Change From Baseline in Bilirubin and Creatinine at Day 8 in Participants Without Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who did not receive the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: micromole per liter (µmol/L)
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 4 | 3
micromole per liter (µmol/L)
  Bilirubin : Baseline | 8.3 (4.43) | 7.7 (4.73)
  Bilirubin : Change at Day 8 | 2.3 (1.71) | -0.3 (2.52)
  Creatinine : Baseline | 79.0 (15.87) | 66.3 (14.36)
  Creatinine : Change at Day 8 | 4.5 (7.72) | -3.7 (3.79)

23. Primary Outcome: Change From Baseline in Bilirubin and Creatinine at Day 8 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
µmol/L
  Bilirubin : Baseline | 7.0 (2.68) | 9.0 (3.56)
  Bilirubin : Change at Day 8 | 0.3 (1.75) | 1.5 (2.08)
  Creatinine : Baseline | 66.8 (13.41) | 69.3 (23.41)
  Creatinine : Change at Day 8 | 3.5 (2.26) | -3.3 (6.65)

24. Primary Outcome: Change From Baseline in Bilirubin and Creatinine at Day 120 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 120
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
µmol/L
  Bilirubin : Baseline | 7.0 (2.68) | 9.0 (3.56)
  Bilirubin : Change at Day 120 | 0.2 (2.56) | -1.0 (3.46)
  Creatinine : Baseline | 66.8 (13.41) | 69.3 (23.41)
  Creatinine : Change at Day 120 | 2.7 (8.87) | -3.8 (8.66)

25. Primary Outcome: Change From Baseline in Bilirubin and Creatinine at Day 8 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 8
Population: Participants in SAF population from Cohorts 3, 4, and 6 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
µmol/L
  Bilirubin : Baseline | 8.2 (3.16) | 7.6 (3.06) | 19.3 (14.74)
  Bilirubin : Change at Day 8 | -0.8 (2.57) | 0.3 (1.64) | -8.0 (9.85)
  Creatinine : Baseline | 66.6 (16.15) | 63.7 (14.94) | 61.3 (5.86)
  Creatinine : Change at Day 8: number analyzed (Participants) | 10 | 9 | 3
  Creatinine : Change at Day 8 | 3.7 (4.42) | 0.8 (2.95) | -2.0 (4.00)

26. Primary Outcome: Change From Baseline in Bilirubin and Creatinine at Day 37 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 37
Population: Participants in SAF population from Cohorts 3, 4, and 6 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
µmol/L
  Bilirubin : Baseline | 8.2 (3.16) | 7.6 (3.06) | 19.3 (14.74)
  Bilirubin : Change at Day 37: number analyzed (Participants) | 10 | 10 | 2
  Bilirubin : Change at Day 37 | -1.2 (2.30) | -0.4 (2.07) | -4.0 (0.00)
  Creatinine : Baseline | 66.6 (16.15) | 63.7 (14.94) | 61.3 (5.86)
  Creatinine : Change at Day 37 | 5.2 (6.53) | -1.2 (4.39) | 1.7 (5.51)

27. Primary Outcome: Change From Baseline in Creatine Kinase at Day 8 in Participants Without Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who did not receive the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: microkatal per liter (μkat/L)
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 4 | 3
microkatal per liter (μkat/L)
  Creatine Kinase : Baseline | 1.3083 (0.3869) | 1.1056 (0.5453)
  Creatine Kinase : Change at Day 8 | -0.2083 (0.1680) | -0.3556 (0.3417)

28. Primary Outcome: Change From Baseline in Creatine Kinase at Day 8 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
μkat/L
  Creatine Kinase : Baseline | 1.2917 (0.5212) | 1.4708 (0.6065)
  Creatine Kinase : Change at Day 8 | -0.1417 (0.2736) | -0.2458 (0.2002)

29. Primary Outcome: Change From Baseline in Creatine Kinase at Day 120 in Participants With Booster Dose (Cohorts 1 and 2)
Time Frame: Baseline, Day 120
Population: Participants in the SAF population from Cohorts 1 and 2 who received the booster dose were analyzed.
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine)
Number analyzed (Participants) | 6 | 4
μkat/L
  Creatine Kinase : Baseline | 1.2917 (0.5212) | 1.4708 (0.6065)
  Creatine Kinase : Change at Day 120 | 0.0750 (0.5691) | -0.5625 (0.2640)

30. Primary Outcome: Change From Baseline in Creatine Kinase at Day 8 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 8
Population: Participants in the SAF population from Cohorts 3, 4 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
μkat/L
  Creatine Kinase : Baseline | 2.2217 (1.0841) | 1.9067 (0.7348) | 1.8056 (0.7473)
  Creatine Kinase : Change at Day 8 | -0.4833 (0.5619) | -0.1217 (0.4350) | -0.4444 (0.4703)

31. Primary Outcome: Change From Baseline in Creatine Kinase at Day 37 in Cohorts 3, 4, and 6
Time Frame: Baseline, Day 37
Population: Participants in the SAF population from Cohorts 3, 4 and 6 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 10 | 3
μkat/L
  Creatine Kinase : Baseline | 2.2217 (1.0841) | 1.9067 (0.7348) | 1.8056 (0.7473)
  Creatine Kinase : Change at Day 37: number analyzed (Participants) | 10 | 10 | 2
  Creatine Kinase : Change at Day 37 | -0.4217 (0.6258) | -0.3583 (0.4508) | -0.4417 (0.1532)

32. Primary Outcome: Number of Participants With Treatment-emergent Serious AEs (SAEs), AE of Special Interest (AESIs) Including Potentially Immune-mediated Medical Conditions (PIMMCs), Medically Attended AEs (MAAEs), and New Onset Chronic Medical Conditions (NOCMCs)
Description: An AE or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, with or without a causal relationship with the vaccine. A TEAE was defined as any event not observed before the first vaccination or any event observed before the first vaccination that worsens in intensity or frequency after exposure. A treatment-emergent SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. Adverse events of special interest were serologically or virologically confirmed SARS-CoV-2 infection or severe COVID-19, NOCMCs, MAAE (hospitalization, an emergency room visit or an otherwise unscheduled visit to or from medical personnel for any reason), and PIMMCs.
Time Frame: Day 1 Up to 16 months
Population: SAF population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
Participants
  SAEs | 2 | 1 | 0 | 2 | 0
  All AESIs | 9 | 6 | 9 | 9 | 3
  MAAEs | 6 | 5 | 5 | 8 | 2
  Severe COVID-19 | 0 | 0 | 0 | 0 | 0
  PIMMCs | 1 | 0 | 0 | 0 | 0
  NOCMCs | 5 | 3 | 2 | 3 | 1
  Serologically or Virologically Confirmed Relevant to COVID-19 | 7 | 6 | 7 | 2 | 2

33. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig)G Level (Spike Wild Type [WT] Variant)
Description: Sera were analyzed for Spike (WT variant)-specific IgG levels pre and post administration of GRT-R910 via enzyme-linked immunosorbent assay (ELISA) and reported as ELISA laboratory units (ELU)/mL (amount of antibodies in the sample according to the unit assigned by the standard).
Time Frame: Baseline, Days 15, 29, 57, 58, 86, 113, 142, 180, 209, 293, 365, 394, 478
Population: Immunogenicity analysis population included participants who received assigned dose(s) at baseline and had at least one available assessment at post-baseline. Participants with available data were analyzed. Data from timepoints collected after reported COVID-19 diagnosis or receipt of external vaccine were excluded.
Measure: Mean (Standard Deviation); unit: ELU/mL
Groups:
- Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine): Healthy participants of age ≥18 to ≤59 years received two doses (Day 1 and Day 29) of GRT-R910 10 μg (homologous prime-boost), at least 2 months after receiving mRNA-based COVID-19 (Pfizer/BioNTech, Moderna) primary series vaccine. Participants were followed for 13 months.
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
ELU/mL
  Baseline | 1472.7 (2054.30) | 927.4 (1432.97) | 8154.3 (10615.60) | 16841.9 (25813.96) | 14127.5 (12307.51)
  Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Change at Day 15 |  |  | 127.6 (187.31) | 2172.0 (5047.29) | -1710.6 (4374.86)
  Change at Day 29: number analyzed (Participants) | 10 | 7 | 8 | 9 | 3
  Change at Day 29 | 11895.9 (13649.88) | 18911.4 (33885.50) | 12487.0 (32915.21) | 6894.5 (10642.03) | -811.4 (4591.85)
  Change at Day 57: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0
  Change at Day 57 | 13611.5 (15451.74) | 18389.1 (32185.66) |  |  |
  Change at Day 58: number analyzed (Participants) | 0 | 0 | 6 | 7 | 3
  Change at Day 58 |  |  | 26631.5 (40900.86) | 20522.6 (23369.31) | 2764.7 (4119.63)
  Change at Day 86: number analyzed (Participants) | 0 | 0 | 6 | 7 | 3
  Change at Day 86 |  |  | 19988.1 (29698.91) | 19290.2 (29851.34) | 3598.0 (4584.89)
  Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Change at Day 113 | 5338.6 (2788.22) | 4429.0 (4194.22) |  |  |
  Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Change at Day 142 | 9912.1 (3698.76) | 4325.1 (998.99) |  |  |
  Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Change at Day 180 | 5617.7 (3997.75) | 43597.9 |  |  |
  Change at Day 209: number analyzed (Participants) | 0 | 0 | 3 | 6 | 1
  Change at Day 209 |  |  | 19612.2 (25727.45) | 13302.7 (35861.57) | 669.2
  Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Change at Day 293 | 8168.6 (1102.84) | 1550.2 |  |  |
  Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Change at Day 365 | 6717.5 |  |  |  |
  Change at Day 394: number analyzed (Participants) | 0 | 0 | 2 | 6 | 1
  Change at Day 394 |  |  | 29156.7 (34271.63) | 19892.7 (29538.44) | -2550.5
  Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Change at Day 478 | 6280.8 | 1787.8 |  |  |

34. Secondary Outcome: Change From Baseline in Neutralizing Antibody (nAb) Levels
Description: Neutralizing antibody titers against live virus were assessed via microneutralization assay. Neutralizing antibody levels were measured for the following variants: WT, Alpha, Beta, Delta, Gamma.
Time Frame: For WT: Baseline, Days 15, 29, 57, 58, 86, 113, 142, 180, 209 293, 365, 394, 478; For Alpha, Beta, Delta, Gamma:Baseline, Days 15, 29, 57, 58, 86, 113, 142, 180, 209 293, 365, 394
Population: Participants in immunogenicity analysis population with available data were analyzed. Data from timepoints collected after reported COVID-19 diagnosis or receipt of external vaccine were excluded.
Measure: Mean (Standard Deviation); unit: titers
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 10 | 10 | 3
titers
  Spike WT Variant : Baseline | 389.3 (648.63) | 364.1 (531.95) | 1598.8 (1614.15) | 1770.6 (2197.25) | 2876.3 (2313.05)
  Spike WT Variant : Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Spike WT Variant : Change at Day 15 |  |  | -181.5 (150.61) | 1291.3 (943.07) | 886.0 (751.13)
  Spike WT Variant : Change at Day 29: number analyzed (Participants) | 10 | 7 | 8 | 9 | 3
  Spike WT Variant : Change at Day 29 | 2736.7 (2296.58) | 5698.4 (8043.68) | 7199.6 (20163.93) | 1520.0 (1481.62) | 403.0 (492.63)
  Spike WT Variant : Change at Day 57: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0
  Spike WT Variant : Change at Day 57 | 3069.6 (3084.54) | 6195.9 (11607.01) |  |  |
  Spike WT Variant : Change at Day 58: number analyzed (Participants) | 0 | 0 | 6 | 7 | 3
  Spike WT Variant : Change at Day 58 |  |  | 27494.5 (60940.14) | 11316.4 (15472.50) | 1684.3 (1330.26)
  Spike WT Variant : Change at Day 86: number analyzed (Participants) | 0 | 0 | 6 | 7 | 3
  Spike WT Variant : Change at Day 86 |  |  | 12417.2 (28027.00) | 9031.7 (9679.50) | 1252.7 (1158.66)
  Spike WT Variant : Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Spike WT Variant : Change at Day 113 | 1877.0 (1083.54) | 1273.0 (998.27) |  |  |
  Spike WT Variant : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Spike WT Variant : Change at Day 142 | 3933.0 (2349.21) | 1479.0 (804.08) |  |  |
  Spike WT Variant : Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike WT Variant : Change at Day 180 | 2722.7 (2504.27) | 11020.0 |  |  |
  Spike WT Variant : Change at Day 209: number analyzed (Participants) | 0 | 0 | 3 | 6 | 1
  Spike WT Variant : Change at Day 209 |  |  | 1896.3 (1539.0) | 4046.8 (4136.43) | 3767.0
  Spike WT Variant : Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike WT Variant : Change at Day 293 | 2527.3 (1758.06) | 412.0 |  |  |
  Spike WT Variant : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike WT Variant : Change at Day 365 | 469.0 |  |  |  |
  Spike WT Variant : Change at Day 394: number analyzed (Participants) | 0 | 0 | 2 | 6 | 1
  Spike WT Variant : Change at Day 394 |  |  | 5771.5 (6639.03) | 6617.8 (8217.53) | 9904.0
  Spike WT Variant : Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike WT Variant : Change at Day 478 | 1059.0 | 163.0 |  |  |
  Spike Alpha Variant : Baseline: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Alpha Variant : Baseline | 212.2 (321.43) | 145.8 (199.14) | 472.5 (318.83) | 2888.6 (3326.23) | 2131.3 (1220.58)
  Spike Alpha Variant : Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Spike Alpha Variant : Change at Day 15 |  |  | 151.0 (4.24) | -473.3 (2492.24) | 462.3 (670.00)
  Spike Alpha Variant : Change at Day 29: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Alpha Variant : Change at Day 29 | 2015.5 (1970.93) | 5750.8 (11303.79) | 5824.3 (10927.20) | 508.2 (2193.32) | 492.7 (169.21)
  Spike Alpha Variant : Change at Day 57: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 57 | 1791.3 (1761.22) | 11060.3 (25154.49) |  |  |
  Spike Alpha Variant : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Alpha Variant : Change at Day 58 |  |  | 10524.0 (15090.23) | 1534.0 (1431.72) | 962.7 (829.00)
  Spike Alpha Variant : Change at Day 86: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Alpha Variant : Change at Day 86 |  |  | 12548.7 (16593.11) | 2793.7 (1513.65) | 6464.3 (6400.08)
  Spike Alpha Variant : Change at Day 113: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 113 | 742.0 (435.92) | 690.7 (501.34) |  |  |
  Spike Alpha Variant : Change at Day 142: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 142 | 1222.0 (341.83) | 647.0 (381.84) |  |  |
  Spike Alpha Variant : Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 180 | 700.3 (1330.07) | 9089.0 |  |  |
  Spike Alpha Variant : Change at Day 209: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Alpha Variant : Change at Day 209 |  |  | 9643.0 | 906.0 (419.01) | 8843.0
  Spike Alpha Variant : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 293 | 1282.0 (944.69) |  |  |  |
  Spike Alpha Variant : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike Alpha Variant : Change at Day 365 | 758.0 |  |  |  |
  Spike Alpha Variant : Change at Day 394: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Alpha Variant : Change at Day 394 |  |  | 2430.0 | 3497.0 (4154.15) | 1441.0
  Spike Beta Variant : Baseline: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Beta Variant : Baseline | 46.8 (24.53) | 54.8 (58.38) | 3049.0 (5611.44) | 728.2 (714.93) | 692.7 (333.52)
  Spike Beta Variant : Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Spike Beta Variant : Change at Day 15 |  |  | 241.0 (101.82) | 1325.3 (1151.95) | 670.0 (323.30)
  Spike Beta Variant : Change at Day 29: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Beta Variant : Change at Day 29 | 620.2 (359.53) | 1645.0 (2331.97) | 946.0 (1918.04) | 438.0 (923.19) | 120.7 (298.41)
  Spike Beta Variant : Change at Day 57: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 57 | 938.2 (483.10) | 1651.0 (2729.72) |  |  |
  Spike Beta Variant : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Beta Variant : Change at Day 58 |  |  | 491.0 (480.77) | 908.7 (725.16) | 355.0 (499.88)
  Spike Beta Variant : Change at Day 86: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Beta Variant : Change at Day 86 |  |  | 551.3 (242.88) | 1479.3 (2024.13) | 1535.0 (1004.73)
  Spike Beta Variant : Change at Day 113: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 113 | 541.0 (442.36) | 531.0 (255.69) |  |  |
  Spike Beta Variant : Change at Day 142: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 142 | 599.3 (426.48) | 608.0 (445.48) |  |  |
  Spike Beta Variant : Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 180 | 473.0 (187.93) | 4357.0 |  |  |
  Spike Beta Variant : Change at Day 209: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Beta Variant : Change at Day 209 |  |  | 59.0 | 474.7 (799.09) | 396.0
  Spike Beta Variant : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 293 | 360.0 (77.78) |  |  |  |
  Spike Beta Variant : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike Beta Variant : Change at Day 365 | 353.0 |  |  |  |
  Spike Beta Variant : Change at Day 394: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Beta Variant : Change at Day 394 |  |  | 29.0 | 2556.0 (2736.07) | 204.0
  Spike Delta Variant : Baseline: number analyzed (Participants) | 6 | 6 | 5 | 5 | 3
  Spike Delta Variant : Baseline | 30.7 (20.15) | 130.8 (287.88) | 204.6 (89.47) | 939.4 (1439.18) | 1111.3 (817.14)
  Spike Delta Variant : Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Spike Delta Variant : Change at Day 15 |  |  | 66.5 (72.83) | 556.0 (903.70) | 35.7 (169.21)
  Spike Delta Variant : Change at Day 29: number analyzed (Participants) | 6 | 6 | 5 | 5 | 3
  Spike Delta Variant : Change at Day 29 | 881.7 (463.61) | 2620.2 (4221.31) | 2190.8 (4501.32) | 441.2 (598.52) | 72.0 (263.90)
  Spike Delta Variant : Change at Day 57: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 57 | 1346.5 (1108.33) | 3149.2 (6124.92) |  |  |
  Spike Delta Variant : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 3 | 3
  Spike Delta Variant : Change at Day 58 |  |  | 5775.0 (10376.28) | 1591.0 (1515.13) | 202.7 (76.05)
  Spike Delta Variant : Change at Day 86: number analyzed (Participants) | 0 | 0 | 4 | 3 | 3
  Spike Delta Variant : Change at Day 86 |  |  | 2020.5 (2913.95) | 861.0 (1075.02) | 1040.7 (1058.26)
  Spike Delta Variant : Change at Day 113: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 113 | 505.0 (364.87) | 455.0 (232.27) |  |  |
  Spike Delta Variant : Change at Day 142: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 142 | 743.3 (455.08) | 312.5 (26.16) |  |  |
  Spike Delta Variant : Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 180 | 543.0 (332.50) | 8896.0 |  |  |
  Spike Delta Variant : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1
  Spike Delta Variant : Change at Day 209 |  |  | 859.5 (211.42) | 463.0 (1029.03) | 2272.0
  Spike Delta Variant : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 293 | 359.5 (6.36) |  |  |  |
  Spike Delta Variant : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike Delta Variant : Change at Day 365 | 361.0 |  |  |  |
  Spike Delta Variant : Change at Day 394: number analyzed (Participants) | 0 | 0 | 2 | 3 | 1
  Spike Delta Variant : Change at Day 394 |  |  | 1478.5 (437.70) | 2093.7 (2175.41) | 2571.0
  Spike Gamma Variant : Baseline: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Gamma Variant : Baseline | 42.2 (19.02) | 64.8 (118.26) | 751.8 (638.95) | 1823.0 (2042.95) | 1387.7 (836.53)
  Spike Gamma Variant : Change at Day 15: number analyzed (Participants) | 0 | 0 | 2 | 3 | 3
  Spike Gamma Variant : Change at Day 15 |  |  | 4.0 (230.52) | 383.3 (577.54) | 30.3 (277.62)
  Spike Gamma Variant : Change at Day 29: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  Spike Gamma Variant : Change at Day 29 | 1595.7 (1258.32) | 2597.3 (4419.00) | 6524.3 (12990.41) | 643.8 (722.95) | 668.7 (654.71)
  Spike Gamma Variant : Change at Day 57: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 57 | 1824.8 (1702.96) | 3001.5 (5634.38) |  |  |
  Spike Gamma Variant : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Gamma Variant : Change at Day 58 |  |  | 12835.0 (21500.00) | 2440.7 (1763.62) | 549.7 (905.99)
  Spike Gamma Variant : Change at Day 86: number analyzed (Participants) | 0 | 0 | 3 | 3 | 3
  Spike Gamma Variant : Change at Day 86 |  |  | 5854.3 (9508.49) | 1361.3 (1933.56) | 633.0 (405.82)
  Spike Gamma Variant : Change at Day 113: number analyzed (Participants) | 3 | 3 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 113 | 568.3 (432.60) | 683.7 (466.31) |  |  |
  Spike Gamma Variant : Change at Day 142: number analyzed (Participants) | 3 | 2 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 142 | 979.7 (1110.39) | 610.0 (571.34) |  |  |
  Spike Gamma Variant : Change at Day 180: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 180 | 1110.0 (732.28) | 4826.0 |  |  |
  Spike Gamma Variant : Change at Day 209: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Gamma Variant : Change at Day 209 |  |  | 394.0 | -295.7 (1059.91) | -103.0
  Spike Gamma Variant : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 293 | 774.0 (15.56) |  |  |  |
  Spike Gamma Variant : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike Gamma Variant : Change at Day 365 | 508.0 |  |  |  |
  Spike Gamma Variant : Change at Day 394: number analyzed (Participants) | 0 | 0 | 1 | 3 | 1
  Spike Gamma Variant : Change at Day 394 |  |  | 310.0 | 1800.3 (3177.44) | -428.0

35. Secondary Outcome: Number of Participants With Immunogenicity Response by Spike IgG and nAb Variants
Description: Immunogenicity response defined as >= 2-fold change in the levels from baseline. Response rate was assessed by Spike IgG wild type and nAb Variants [wild type, alpha, beta, gamma, delta]. Number of participants with immunogenicity response at any post-baseline timepoint are provided.
Time Frame: Baseline to 478 days
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 10 | 7 | 8 | 9 | 3
Participants
  IgG WT | 9 | 6 | 5 | 4 | 0
  nAb WT | 9 | 5 | 4 | 5 | 1
  nAb Alpha: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  nAb Alpha | 5 | 5 | 2 | 1 | 2
  nAb Beta: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  nAb Beta | 6 | 5 | 1 | 3 | 1
  nAb Delta: number analyzed (Participants) | 6 | 5 | 5 | 5 | 3
  nAb Delta | 6 | 4 | 4 | 1 | 1
  nAb Gamma: number analyzed (Participants) | 6 | 6 | 4 | 5 | 3
  nAb Gamma | 6 | 5 | 2 | 0 | 0

36. Secondary Outcome: Change From Baseline in T Cell Response by Spike Pools (ex Vivo ELISpot)
Description: Peripheral blood mononuclear cells (PBMCs) were isolated from whole blood. T cell responses to SARS-CoV-2 D614G were assessed via ex vivo IFNγ ELISpot assay (methods). Cells were stimulated with overlapping peptide (OLP) pools containing peptides that were 15 amino acids in length (15mers) and spanning both S subunits (Spike pool 1-2, 3-4 [S1], 5-6, and 7-8 [S2]).
Time Frame: Baseline, Days 8, 29, 58, 113, 142, 180, 209, 293, 365, 478
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Spot Forming Unit (SFU) per 10^6 cells
Groups:
- Cohort 1: GRT-R910 10 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine): Healthy participants of age ≥60 years received prime dose (on Day 1) of GRT-R910 10 μg intramuscularly at least 2 months after receiving a first-generation COVID-19 (AstraZeneca) vaccine primary series. A subset of participants elected to receive a booster vaccination of GRT-R910 10 μg which was administered 113 days after the prime vaccination. Participants not receiving booster dose were followed for 12 months, and participants receiving booster dose were followed for 16 months.
- Cohort 2: GRT-R910 30 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine): Healthy participants of age ≥60 years received prime dose (on Day 1) of GRT-R910 30 μg intramuscularly at least 2 months after receiving a first-generation COVID-19 (AstraZeneca) vaccine primary series. A subset of participants elected to receive a booster vaccination of GRT-R910 10 μg, which was administered 113 days after the prime vaccination. Participants not receiving booster dose were followed for 12 months, and participants receiving booster dose were followed for 16 months.
- Cohort 3: GRT-R910 10 μg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine): Healthy participants of age ≥60 years received two doses (Day 1 and Day 29) of GRT-R910 10 μg (homologous prime-boost), at least 2 months after receiving an adenoviral COVID-19 (AstraZeneca, Janssen) primary series vaccine. Participants were followed for 13 months.
- Cohort 4: GRT-R910 10 μg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine): Healthy participants of age ≥60 years received two doses (Day 1 and Day 29) of GRT-R910 10 μg (homologous prime-boost), at least 2 months after receiving a messenger ribonucleic acid (mRNA)-based COVID-19 (Pfizer/ BioNTech, Moderna) primary series vaccine. Participants were followed for 13 months.
- Cohort 6: GRT-R910 10 μg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine): Healthy participants of age ≥18 to ≤59 years received two doses (Day 1 and Day 29) of GRT-R910 10 μg (homologous prime-boost), at least 2 months after receiving mRNA-based COVID-19 (Pfizer/BioNTech, Moderna) primary series vaccine. Participants were followed for 13 months.
Arm/Group | Cohort 1: GRT-R910 10 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 μg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 μg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 μg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 9 | 7 | 8 | 6 | 1
Spot Forming Unit (SFU) per 10^6 cells
  Spike pool 1_2 : Baseline | 62.5 (61.35) | 62.5 (53.93) | 75.0 (82.22) | 17.9 (7.14) | 15.0
  Spike pool 1_2 : Change at Day 8 | -5.0 (41.06) | -5.7 (31.38) | -19.4 (30.81) | -0.4 (1.02) | 0.0
  Spike pool 1_2 : Change at Day 29: number analyzed (Participants) | 9 | 7 | 6 | 5 | 1
  Spike pool 1_2 : Change at Day 29 | 46.7 (119.95) | 20.7 (37.10) | 30.0 (46.61) | 1.5 (3.35) | 0.0
  Spike pool 1_2 : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 1
  Spike pool 1_2 : Change at Day 58 |  |  | 29.4 (34.60) | 9.5 (15.25) | 0.0
  Spike pool 1_2 : Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 113 | -0.8 (37.10) | 1.3 (38.65) |  |  |
  Spike pool 1_2 : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 142 | -13.8 (33.61) | 6.7 (11.55) |  |  |
  Spike pool 1_2 : Change at Day 180: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 180 | 1.3 (40.66) | 30.0 |  |  |
  Spike pool 1_2 : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  Spike pool 1_2 : Change at Day 209 |  |  | 52.5 (84.85) | 7.5 (12.99) |
  Spike pool 1_2 : Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 293 | -2.5 (33.63) | 40.0 |  |  |
  Spike pool 1_2 : Change at Day 365: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 365 | 40.0 |  |  |  |
  Spike pool 1_2 : Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 1_2 : Change at Day 478 | 20.0 | 82.5 |  |  |
  Spike pool 3_4 : Baseline: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 3_4 : Baseline | 30.9 (19.86) | 51.1 (37.16) | 69.7 (56.35) | 94.6 (180.45) | 15.0
  Spike pool 3_4 : Change at Day 8: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 3_4 : Change at Day 8 | 10.3 (27.79) | 10.4 (23.25) | 5.9 (27.35) | -22.5 (41.35) | 0.0
  Spike pool 3_4 : Change at Day 29: number analyzed (Participants) | 8 | 7 | 6 | 4 | 1
  Spike pool 3_4 : Change at Day 29 | 24.1 (38.52) | 16.1 (31.72) | 34.2 (52.65) | 21.3 (47.63) | 0.0
  Spike pool 3_4 : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 1
  Spike pool 3_4 : Change at Day 58 |  |  | 23.8 (29.26) | 2.0 (9.25) | 0.0
  Spike pool 3_4 : Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 113 | 4.6 (22.16) | -15.0 (36.97) |  |  |
  Spike pool 3_4 : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 142 | 14.2 (53.70) | -25.0 (43.30) |  |  |
  Spike pool 3_4 : Change at Day 180: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 180 | 0.0 | 62.5 |  |  |
  Spike pool 3_4 : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  Spike pool 3_4 : Change at Day 209 |  |  | 61.3 (76.01) | -17.5 (30.31) |
  Spike pool 3_4 : Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 293 | 58.3 (92.68) | 0.0 |  |  |
  Spike pool 3_4 : Change at Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 3_4 : Change at Day 478 | 225.0 | 0.0 |  |  |
  Spike pool 5_6 : Baseline: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 5_6 : Baseline | 34.4 (32.37) | 33.9 (40.51) | 37.2 (41.18) | 34.6 (29.34) | 15.0
  Spike pool 5_6 : Change at Day 8: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 5_6 : Change at Day 8 | 11.6 (37.03) | 11.4 (32.56) | 3.4 (20.09) | -4.6 (11.23) | 0.0
  Spike pool 5_6 : Change at Day 29: number analyzed (Participants) | 8 | 7 | 6 | 4 | 1
  Spike pool 5_6 : Change at Day 29 | 17.5 (68.54) | 9.6 (25.31) | 36.7 (36.11) | 23.1 (36.93) | 0.0
  Spike pool 5_6 : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 1
  Spike pool 5_6 : Change at Day 58 |  |  | 62.5 (45.55) | -3.0 (4.47) | 0.0
  Spike pool 5_6 : Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 113 | -7.5 (17.18) | 0.0 (0.00) |  |  |
  Spike pool 5_6 : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 142 | -5.4 (25.02) | 17.5 (30.31) |  |  |
  Spike pool 5_6 : Change at Day 180: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 180 | 0.0 | 25.0 |  |  |
  Spike pool 5_6 : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  Spike pool 5_6 : Change at Day 209 |  |  | 75.0 (106.07) | -10.0 (10.00) |
  Spike pool 5_6 : Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 293 | 5.8 (19.42) | 32.5 |  |  |
  Spike pool 5_6 : Change at Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 5_6 : Change at Day 478 | 15.0 | 67.5 |  |  |
  Spike pool 7_8 : Baseline: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 7_8 : Baseline | 20.9 (6.94) | 25.7 (13.13) | 30.9 (22.83) | 16.3 (3.06) | 15.0
  Spike pool 7_8 : Change at Day 8: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike pool 7_8 : Change at Day 8 | 3.4 (9.54) | 52.1 (88.04) | -11.6 (17.27) | -1.3 (3.06) | 0.0
  Spike pool 7_8 : Change at Day 29: number analyzed (Participants) | 8 | 7 | 6 | 4 | 1
  Spike pool 7_8 : Change at Day 29 | 8.4 (23.37) | 80.4 (148.42) | 9.2 (29.18) | -1.9 (3.75) | 0.0
  Spike pool 7_8 : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 1
  Spike pool 7_8 : Change at Day 58 |  |  | 8.8 (17.50) | -1.5 (3.35) | 0.0
  Spike pool 7_8 : Change at Day 113: number analyzed (Participants) | 6 | 4 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 113 | -0.8 (11.58) | 15.0 (42.62) |  |  |
  Spike pool 7_8 : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 142 | 0.0 (15.25) | 169.2 (308.28) |  |  |
  Spike pool 7_8 : Change at Day 180: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 180 | 0.0 | 20.0 |  |  |
  Spike pool 7_8 : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  Spike pool 7_8 : Change at Day 209 |  |  | 13.8 (19.45) | 1.7 (2.89) |
  Spike pool 7_8 : Change at Day 293: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 293 | 7.5 (9.01) | -32.5 |  |  |
  Spike pool 7_8 : Change at Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 478: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0
  Spike pool 7_8 : Change at Day 478 | 20.0 | 27.5 |  |  |

37. Secondary Outcome: Change From Baseline in T Cell Response by T Cell Epitope (TCE) Pools (ex Vivo ELISpot)
Description: PBMCs were isolated from whole blood. T cell responses to conserved SARS-CoV-2 viral epitopes were assessed via ex vivo IFNγ ELISpot assay (methods). Responses to Nucleocapsid (Nuc) and open reading frame 3a (ORF3a)/Membrane TCE regions were assessed using OLP pools.
Time Frame: Baseline, Days 8, 29, 58, 113, 142, 180, 209, 293, 365, 478
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: SFU per 10^6 cells
Groups:
- Cohort 3: GRT-R910 10 μg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine: Healthy participants of age ≥60 years received two doses (Day 1 and Day 29) of GRT-R910 10 μg (homologous prime-boost), at least 2 months after receiving an adenoviral COVID-19 (AstraZeneca, Janssen) primary series vaccine. Participants were followed for 13 months.
Arm/Group | Cohort 1: GRT-R910 10 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 μg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine | Cohort 4: GRT-R910 10 μg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 μg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 0 | 7 | 8 | 6 | 1
SFU per 10^6 cells
  Nuc OLP : Baseline |  | 15.0 (0.00) | 15.0 (0.00) | 16.3 (3.06) | 15.0
  Nuc OLP : Change at Day 8: number analyzed (Participants) | 0 | 7 | 8 | 5 | 1
  Nuc OLP : Change at Day 8 |  | 3.6 (9.45) | 0.0 (0.00) | -1.5 (3.35) | 0.0
  Nuc OLP : Change at Day 29: number analyzed (Participants) | 0 | 7 | 6 | 4 | 1
  Nuc OLP : Change at Day 29 |  | 1.1 (2.83) | 3.3 (5.40) | 0.0 (0.00) | 0.0
  Nuc OLP : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0
  Nuc OLP : Change at Day 58 |  |  | 3.8 (7.50) | 0.0 (0.00) |
  Nuc OLP : Change at Day 113: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Nuc OLP : Change at Day 113 |  | 0.0 (0.00) |  |  |
  Nuc OLP : Change at Day 142: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Nuc OLP : Change at Day 142 |  | 0.0 (0.00) |  |  |
  Nuc OLP : Change at Day 180: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Nuc OLP : Change at Day 180 |  | 0.0 |  |  |
  Nuc OLP : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  Nuc OLP : Change at Day 209 |  |  | 0.0 (0.00) | 0.0 (0.00) |
  Nuc OLP : Change at Day 293: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Nuc OLP : Change at Day 293 |  | 0.0 |  |  |
  Nuc OLP : Change at Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Nuc OLP : Change at Day 478: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  ORF3a/Membrane OLP : Baseline |  | 17.9 (7.56) | 19.4 (9.04) | 15.0 (0.00) | 15.0
  ORF3a/Membrane OLP : Change at Day 8: number analyzed (Participants) | 0 | 7 | 6 | 5 | 1
  ORF3a/Membrane OLP : Change at Day 8 |  | -0.4 (0.94) | 0.8 (2.04) | 0.0 (0.00) | 0.0
  ORF3a/Membrane OLP : Change at Day 29: number analyzed (Participants) | 0 | 7 | 6 | 4 | 1
  ORF3a/Membrane OLP : Change at Day 29 |  | 15.4 (26.24) | 0.0 (6.32) | 0.0 (0.00) | 0.0
  ORF3a/Membrane OLP : Change at Day 58: number analyzed (Participants) | 0 | 0 | 4 | 5 | 0
  ORF3a/Membrane OLP : Change at Day 58 |  |  | 4.4 (16.12) | 3.5 (7.83) |
  ORF3a/Membrane OLP : Change at Day 113: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  ORF3a/Membrane OLP : Change at Day 113 |  | 0.0 (0.00) |  |  |
  ORF3a/Membrane OLP : Change at Day 142: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  ORF3a/Membrane OLP : Change at Day 142 |  | 0.0 (0.00) |  |  |
  ORF3a/Membrane OLP : Change at Day 180: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ORF3a/Membrane OLP : Change at Day 180 |  | 47.5 |  |  |
  ORF3a/Membrane OLP : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 3 | 0
  ORF3a/Membrane OLP : Change at Day 209 |  |  | 0.0 (0.00) | 0.0 (0.00) |
  ORF3a/Membrane OLP : Change at Day 293: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ORF3a/Membrane OLP : Change at Day 293 |  | 0.0 |  |  |
  ORF3a/Membrane OLP : Change at Day 365: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  ORF3a/Membrane OLP : Change at Day 478: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Change From Baseline in Immunogenicity Response by TCE Pools (in Vitro Stimulation)
Description: PBMCs were isolated from whole blood. T cell responses to conserved SARS-CoV-2 viral epitopes were assessed via IFNγ ELISpot assay following in vitro stimulation. Responses to Nuc, ORF3a, and membrane TCE regions were assessed using OLP pools.
Time Frame: Baseline, Days 8, 29, 58, 113, 142, 180, 209, 293
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: SFU per 10^6 cells
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 7 | 7 | 6 | 6 | 2
SFU per 10^6 cells
  Nuc OLP : Baseline: number analyzed (Participants) | 6 | 7 | 6 | 6 | 2
  Nuc OLP : Baseline | 502.5 (609.64) | 1823.6 (2091.63) | 2292.5 (2198.52) | 2890.0 (3792.10) | 10397.5 (3680.49)
  Nuc OLP : Change at Day 8: number analyzed (Participants) | 6 | 7 | 6 | 6 | 2
  Nuc OLP : Change at Day 8 | -122.5 (637.16) | 353.6 (2385.88) | -1280.8 (2440.97) | 145.8 (669.91) | -4355.0 (6264.97)
  Nuc OLP : Change at Day 29: number analyzed (Participants) | 6 | 6 | 4 | 5 | 2
  Nuc OLP : Change at Day 29 | 206.7 (498.15) | -360.8 (3094.77) | -541.3 (479.69) | 371.0 (2366.67) | -5890.0 (8683.27)
  Nuc OLP : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 4 | 1
  Nuc OLP : Change at Day 58 |  |  | -183.3 (409.95) | 1482.5 (2755.78) | 55.0
  Nuc OLP : Change at Day 113: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Nuc OLP : Change at Day 113 | 1341.7 (1743.64) | 10.0 (748.55) |  |  |
  Nuc OLP : Change at Day 142: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0
  Nuc OLP : Change at Day 142 | 656.7 (772.89) | 655.0 (1079.11) |  |  |
  Nuc OLP : Change at Day 180: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Nuc OLP : Change at Day 180 |  | 140.0 |  |  |
  Nuc OLP : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 2 | 0
  Nuc OLP : Change at Day 209 |  |  | 2487.5 (3744.13) | -615.0 (466.69) |
  Nuc OLP : Change at Day 293: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  Nuc OLP : Change at Day 293 | 315.0 (1154.69) |  |  |  |
  ORF3a OLP : Baseline: number analyzed (Participants) | 7 | 6 | 5 | 4 | 0
  ORF3a OLP : Baseline | 472.1 (485.03) | 695.8 (1328.89) | 364.0 (355.17) | 298.8 (249.21) |
  ORF3a OLP : Change at Day 8: number analyzed (Participants) | 7 | 5 | 5 | 4 | 0
  ORF3a OLP : Change at Day 8 | -125.0 (441.99) | -555.0 (1544.96) | 163.0 (560.80) | 66.3 (101.93) |
  ORF3a OLP : Change at Day 29: number analyzed (Participants) | 7 | 4 | 4 | 4 | 0
  ORF3a OLP : Change at Day 29 | -81.4 (425.82) | 126.3 (259.27) | -86.3 (248.04) | 111.3 (105.39) |
  ORF3a OLP : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 3 | 0
  ORF3a OLP : Change at Day 58 |  |  | -15.0 (232.86) | 155.0 (330.95) |
  ORF3a OLP : Change at Day 113: number analyzed (Participants) | 5 | 1 | 0 | 0 | 0
  ORF3a OLP : Change at Day 113 | 170.0 (604.78) | 0.0 |  |  |
  ORF3a OLP : Change at Day 142: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  ORF3a OLP : Change at Day 142 | 211.0 (446.86) | 68.3 (70.06) |  |  |
  ORF3a OLP : Change at Day 180: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  ORF3a OLP : Change at Day 180 |  | 495.0 |  |  |
  ORF3a OLP : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  ORF3a OLP : Change at Day 209 |  |  | 0.0 (0.00) | -340.0 |
  ORF3a OLP : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  ORF3a OLP : Change at Day 293 | -385.0 (544.47) |  |  |  |
  Membrane OLP : Baseline: number analyzed (Participants) | 7 | 6 | 5 | 4 | 0
  Membrane OLP : Baseline | 993.6 (1190.16) | 347.5 (270.40) | 1277.0 (2005.93) | 645.0 (434.40) |
  Membrane OLP : Change at Day 8: number analyzed (Participants) | 6 | 6 | 5 | 4 | 0
  Membrane OLP : Change at Day 8 | 152.5 (608.04) | 235.8 (1078.42) | 1794.0 (3722.19) | 1846.3 (2972.90) |
  Membrane OLP : Change at Day 29: number analyzed (Participants) | 7 | 4 | 4 | 4 | 0
  Membrane OLP : Change at Day 29 | -95.0 (1336.77) | 1041.3 (882.95) | -190.0 (299.14) | 1290.0 (2321.25) |
  Membrane OLP : Change at Day 58: number analyzed (Participants) | 0 | 0 | 3 | 3 | 0
  Membrane OLP : Change at Day 58 |  |  | 973.3 (848.27) | 2308.3 (4019.82) |
  Membrane OLP : Change at Day 113: number analyzed (Participants) | 5 | 1 | 0 | 0 | 0
  Membrane OLP : Change at Day 113 | 281.0 (1127.42) | 0.0 |  |  |
  Membrane OLP : Change at Day 142: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Membrane OLP : Change at Day 142 | 843.0 (1741.89) | 281.7 (617.70) |  |  |
  Membrane OLP : Change at Day 180: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Membrane OLP : Change at Day 180 |  | 1075.0 |  |  |
  Membrane OLP : Change at Day 209: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  Membrane OLP : Change at Day 209 |  |  | 125.0 (176.78) | -820.0 |
  Membrane OLP : Change at Day 293: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  Membrane OLP : Change at Day 293 | -280.0 (1909.19) |  |  |  |

39. Secondary Outcome: Number of Participants With Immunogenicity Response by Spike Pools and TCE Pools (ex Vivo ELISpot)
Description: T cell responses to SARS-CoV-2 D614G and conserved non-Spike epitopes were assessed via ex vivo IFNγ ELISpot assay (methods) using OLP pools containing peptides that were 15 amino acids in length and spanning both S subunits (Spike pool 1-2, 3-4 [S1], 5-6, and 7-8 [S2]) and TCE regions Nuc and ORF3a/Membrane. Immunogenicity response was defined as >= 2-fold change in levels from baseline. Response rate to both Spike pools (Spike pool 1-2, 3-4, 5-6, and 7-8) and TCE pools (Nuc OLP and ORF3a/Membrane OLP) was assessed.
Time Frame: Baseline to 478 days
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: GRT-R910 10 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 μg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 μg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 μg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 μg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
Number analyzed (Participants) | 9 | 7 | 8 | 6 | 1
Participants
  Spike Pool 1_2 | 4 | 1 | 1 | 2 | 0
  Spike Pool 3_4: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike Pool 3_4 | 4 | 3 | 1 | 0 | 0
  Spike Pool 5_6: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike Pool 5_6 | 3 | 2 | 5 | 1 | 0
  Spike Pool 7_8: number analyzed (Participants) | 8 | 7 | 8 | 6 | 1
  Spike Pool 7_8 | 3 | 5 | 3 | 0 | 0
  TCE Pool : Nuc OLP: number analyzed (Participants) | 0 | 7 | 8 | 6 | 1
  TCE Pool : Nuc OLP |  | 1 | 1 | 0 | 0
  TCE Pool : Mem/ORF3a OLP: number analyzed (Participants) | 0 | 7 | 8 | 6 | 1
  TCE Pool : Mem/ORF3a OLP |  | 2 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose to month 16
Description: The Safety Analysis Population will include all participants who received any dose of GRT-R910. AEs were collected as solicited and unsolicited AEs. The preferred term reported as both solicited and unsolicited AEs are presented under more than one system organ class due to the difference in nature of the events.
Arm/Group | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7 | 0/10 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/7 | 0/10 | 2/10 | 0/3
Other Adverse Events (participants affected / at risk) | 10/10 | 7/7 | 10/10 | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) (N=10) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) (N=7) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) (N=10) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) (N=10) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) (N=3)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: GRT-R910 10 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) (N=10) | Cohort 2: GRT-R910 30 µg, Age ≥60 Years (Receipt of AstraZeneca Vaccine) (N=7) | Cohort 3: GRT-R910 10 µg, ≥60 Years, (Receipt of AstraZeneca or Janssen COVID-19 Vaccine) (N=10) | Cohort 4: GRT-R910 10 µg, ≥60 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) (N=10) | Cohort 6: GRT-R910 10 µg, ≥18 to ≤59 Years, (Receipt of Pfizer/BioNTech, Moderna COVID-19 Vaccine) (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 10 | 7 | 10 | 10 | 3
Fatigue (General disorders) | 6 | 6 | 10 | 8 | 3
Feverish (Chills/Sweating) (General disorders) | 7 | 7 | 9 | 7 | 3
Malaise (General disorders) | 5 | 6 | 10 | 9 | 3
Headache (General disorders) | 8 | 6 | 9 | 4 | 3
Muscle Pain (General disorders) | 4 | 7 | 8 | 5 | 3
Arthralgia (General disorders) | 3 | 6 | 6 | 4 | 2
Nausea or Vomiting (General disorders) | 1 | 4 | 5 | 5 | 2
Injection site swelling (General disorders) | 2 | 4 | 1 | 2 | 2
Fever (General disorders) | 0 | 2 | 2 | 2 | 1
Injection site erythema (General disorders) | 0 | 2 | 3 | 0 | 1
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT05148962/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT05148962/SAP_001.pdf